CLINICAL TRIAL: NCT03484845
Title: Lactoferrin Versus Ferrous Fumarate for Treatment of Mild to Moderate Iron Deficiency Anemia During Pregnancy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amaal Khalil Hamed, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: u1111-1210-1436
Record Dates: First submitted 2018-03-20; First posted 2018-04-02 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Iron Deficiency Anemia of Pregnancy
MeSH Terms: interventions — Lactoferrin; ferrous fumarate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral lactoferrin (Active Comparator): women who take oral lactoferrin sachets 100 mg twice daily for one month.
  Interventions: Drug: Lactoferrin and ferrous fumarate
- Oral ferrous fumarate (Active Comparator): women who take oral ferrous fumarate tablet 30 mg elemental iron twice daily for one month.
  Interventions: Drug: Lactoferrin and ferrous fumarate
- Combined lactoferrin & ferrous fumarate (Active Comparator): women who take lactoferrin sachets 100 mg and ferrous fumarate tablet 30 mg elemental iron once daily for one month.
  Interventions: Drug: Lactoferrin and ferrous fumarate

INTERVENTIONS:
Drug: Lactoferrin and ferrous fumarate — * Group 1:include 50 women will receive oral lactoferrin 100mg twice daily .
  * Group 2: include 50 women will receive oral Ferrous fumarate 30mg elemental iron twice daily .
  * Group 3: include 50 women will receive oral combined lactoferrin 200mg and ferrous fumarate 60mg elemental iron once daily .
  Other Names: pravotin sachets and vitayami tablets

SUMMARY:
This study will conducted to evaluate and comparison between the effectiveness, safety and acceptability of lactoferrin alone, ferrous fumarate alone and combination of both for the treatment of mild to moderate IDA during pregnancy.

DETAILED DESCRIPTION:
Anemia in pregnancy is a major public health problem, where it has been estimated that 41.8% of pregnant women worldwide are anemic .

Iron deficiency anemia (IDA) is the condition in which there is anemia due to a lack of iron. IDA develops when available iron is insufficient to support normal red cell production and is the most common type of anemia Anemia has a significant impact on the health of the fetus as well as that of the mother. It impairs the oxygen delivery through the placenta to the fetus and interferes with the normal intrauterine growth, leading to fetal loss and perinatal deaths. Anemia is associated with increased preterm labor (28.2%), preeclampsia (31.2%), and maternal sepsis.

The daily requirement of iron is around 1.5 mg in nonpregnant women. This requirement increases dramatically during pregnancy to reach 6-7 mg/day (total 1000 mg) with advanced gestational age. Pregnancy causes a twofold to threefold increase in the requirement for iron and a 10- to 20-fold increase in folate requirement. The increase in demand for iron is mainly due to fetal requirement, placenta, blood volume, tissue accretion, and the intra-partum potential for blood loss

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from 24-36 weeks of gestation.
* Mild to moderate anemia.

Exclusion Criteria:

* Women with a history of anemia due to any other causes other than IDA.
* Severe anemia requiring blood transfusion.
* History of peptic ulcer.
* known hypersensitivity to iron preparations.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Increase in blood hemoglobin. | one month
  mean difference in hemoglobin level between pre treatment and post treatment.